CLINICAL TRIAL: NCT04449484
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of MEDI1341 in Subjects With Parkinson's Disease
Brief Title: Multiple Ascending Dose Study of MEDI1341 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6340C00002
Record Dates: First submitted 2019-04-23; First posted 2020-06-26 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Subjects are randomised to one of two groups within a cohort of 12 subjects (N=9 MEDI1341; N=3 Placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI1341 (Experimental): 3 doses given at 4 week intervals
  Interventions: Drug: MEDI1341
- Placebo (Placebo Comparator): 3 doses given at 4 week intervals
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI1341 — Intravenous infusion over 60 minutes
  Other Names: TAK-341
  Arms: MEDI1341
Other: Placebo — Intravenous infusion over 60 minutes
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study of multiple ascending iv doses of MEDI341 in male and female subjects with Parkinson's Disease.

DETAILED DESCRIPTION:
The study will include up to 3 cohorts, with 12 subjects in each, for a total of up to 36 randomised subjects.

The study comprises a screening period of up to 49 days, an 8-week double-blind treatment period, and a 13-week follow-up period. Each subject will receive three 60 minute iv infusions of MEDI1341 or placebo during the 8-week treatment period, with 4 weeks between infusions. The overall study duration (enrolment, treatment, and follow-up periods) will be up to 28 weeks per subject.

A Dose Escalation Committee will review data from each cohort to allow progression to the next higher dose cohort in the study.

ELIGIBILITY:
Inclusion criteria:

1. Subjects must be aged 40 to 85 years, inclusive, on the day of randomization.
2. Meet criteria for a diagnosis of mild-to-moderate idiopathic PD according to the United Kingdom Parkinson's Disease Society Brain Bank criteria (Hughes et al 1992)
3. PD should be stage 1 to 3 using the Hoehn and Yahr scale as modified (Goetz et al 2004).
4. Subjects receiving medications for PD should have been on a stable dosing regimen of their medication(s) for ≥ 1 month before randomization, with no expectation of a need to change the medications or dosing regimen for the duration of the study, barring unforeseen circumstances. (For subjects who are not currently receiving medications to treat PD, there should be no expectation of a need to initiate these for the duration of the study).
5. Subjects must have a body weight of 45 to 120 kg, inclusive, and a body mass index of 18 to 34 kg/m2, inclusive at screening and at check-in for the first infusion.
6. Subjects may be male or female. Female subjects must of non-childbearing potential (postmenopausal and/or surgically sterile.
7. Postmenopausal women must have had ≥ 12 months of spontaneous amenorrhea (with a follicle-stimulating hormone [FSH] concentration ≥ 26 mIU/mL in women ≤ 60 years of age; women > 60 years of age do not require an FSH test) and must have had a negative serum pregnancy test result at screening.

   Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy (oophorectomy), salpingectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure by an operative report, ultrasound, or other verifiable medical documentation.
8. Men who are biologically capable of fathering children must agree and commit to use an adequate form of double-barrier contraception for the duration of the treatment period and for 5 half lives (100 days) after the last administration of study intervention. A male subject is considered capable of fathering children even if his sexual partner is sterile or using contraceptives.

   Men who are biologically capable of fathering children must also agree to refrain from sperm donation for the duration of the treatment period and for 5 half-lives or 90 days (whichever is longer) after the last administration of study intervention.
9. Subjects must, in the investigator's opinion, understand the nature of the study and must provide signed and dated written informed consent before the conduct of any study-related procedures.
10. Subjects must, in the opinion of the investigator, be able to participate in all scheduled evaluations, likely to be compliant, and likely to complete all required tests, including magnetic resonance imaging (MRI) brain scans and lumbar punctures (LPs). (Note: The investigator should assess the physical and functional needs of the subject at screening, as participation in the study may be contingent upon the availability and willingness of a caregiver to attend with the subject at all study visits.)
11. Subjects must be able to read, write, and speak fluently in English and/or Spanish.
12. Subjects must agree not to post any personal medical data related to the study or information related to the study on any website or social media site (eg, Facebook, Twitter, Instagram, etc) until the study has been completed.
13. Subjects must have a MoCA total score of ≥ 24.

Exclusion Criteria:

1. In the opinion of the investigator, a recent clinically significant illness (other than PD), infection, medical/surgical procedure, or significant trauma within 30 days prior to screening, or between screening and randomization, that is likely to deteriorate, compromise the subject's safety or ability to complete the study, or compromise the interpretation of the study results (Note: a history of coronavirus disease 2019 [COVID 19] infection with unresolved medical sequelae would be considered exclusionary.)
2. Presence of a serious or unstable clinically significant illness, including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic or autoimmune disease (eg, multiple sclerosis), hematologic or other major disease, which, in the judgment of the investigator, is poorly controlled or otherwise likely to deteriorate, compromise the subject's safety or ability to complete the study, or compromise the interpretation of the study results
3. Significant neurological disease affecting the CNS (other than PD) that, in the opinion of the investigator, may affect motor function or the ability to complete the study, including but not limited to progressive supranuclear palsy, multiple system atrophy (MSA; including MSA-P and MSA-C or other MSA terminology: striatonigral degeneration, olivopontocerebellar atrophy or autonomic failure), postencephalitic parkinsonism, metabolic diseases with parkinsonian signs and symptoms (eg, Wilson disease, manganese exposure) or other secondary forms of Parkinsonism, and ischemic or traumatic brain injury (including multiple episodes of head trauma, or head trauma resulting in protracted loss of consciousness within the 5 years prior to screening or between screening and randomization)
4. Brain MRI scan that shows clinically significant evidence of malignant, ischemic, demyelinating, structural, or degenerative brain disease or has findings that compromise the safety of LP
5. Has undergone surgery for the treatment of PD (eg, pallidotomy, deep brain stimulation, fetal tissue transplantation) or has undergone any other brain surgery at any time, even for non-PD conditions
6. History of epilepsy or seizures, except febrile childhood seizures
7. History of transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to screening or between screening and randomization
8. Presence of any psychiatric disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V; APA 2013) or symptom if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of the study results, affect motor function assessment, or affect the subject's ability to complete the study
9. A diagnosis of intellectual disability (intellectual developmental disorder) or mental retardation, or significant inherited cognitive impairment
10. Suicidality, represented by answering "yes" to Question 4 or Question 5 on the C SSRS, indicating active suicidal ideation with any intent to act, during the subject's lifetime, as assessed at screening, or between screening and randomization
11. Suicidal behavior such that a determination of "yes" is made on the Suicidal Behavior section of the C SSRS for "Actual Attempt," "Interrupted Attempt," "Aborted Attempt," or "Preparatory Acts or Behavior," during the subject's lifetime, as assessed at screening, or between screening and randomization
12. History of alcohol or drug abuse or dependence (except nicotine dependence), as defined by the DSM-V, within 2 years prior to screening or between screening and randomization
13. Within 1 year prior to screening, any of the following: myocardial infarction; hospitalization for congestive heart failure; hospitalization for, or symptoms of unstable angina; unexplained syncope
14. Moderate or severe congestive heart failure, or known ejection fraction < 40%
15. Known significant structural heart disease (eg, significant valvular disease, hypertrophic cardiomyopathy) that is considered likely to lead to a deterioration of cardiac function over the course of the study
16. History of cancer within 5 years prior to screening or between screening and randomization, with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin
17. History of allergy/hypersensitivity to immunizations or immunoglobulins
18. Any condition that, in the opinion of the investigator or medical monitor, makes the subject unsuitable for the study
19. Requires treatment with another monoclonal antibody
20. Use of any investigational medicine, device, or biologic within 3 months or 5 half-lives of that intervention (whichever is longer) prior to screening
21. Previous allogeneic bone marrow or stem cell transplant
22. Use of typical or atypical antipsychotic medication, or other medication with dopamine antagonist properties (eg, metoclopramide, domperidone), within 6 months prior to randomization
23. Use of immunosuppressive medication within 6 months prior to randomization. (Note: Inhaled and topical corticosteroids are permitted. Low-dose systemic corticosteroids [< 10 mg per day prednisone or equivalent], for autoimmune disease that is considered to be quiescent, in remission, or otherwise well controlled are permitted). Other immunosuppressive drugs and biologics are contraindicated.
24. Received non-leukocyte depleted whole blood transfusion within 6 months prior to screening
25. Received any commercially available vaccine within 30 days prior to randomization. (Note: for COVID-19 vaccines authorized by the FDA for emergency use, this time frame applies from last vaccination or booster dose, whichever is required to consider vaccination complete in line with applicable guidance.)
26. Participation in another study investigating:

    1. Active or passive immunization against α synuclein for PD, at any time prior to screening, or
    2. Immunoglobulin G therapy within 6 months before screening
27. Any clinically significant abnormality as determined by investigator at screening or between screening and randomization in physical examination, vital signs, ECG, or clinical laboratory test results that may compromise the subject's safety or ability to complete the study or compromise the interpretation of the study results
28. Presence of any of the following MRI contraindications: pacemaker; cardiac defibrillator; spinal cord or vagus nerve stimulator; aneurysm clip; artificial heart valve; recent (within one year) coronary or carotid stent; ear implant; CSF shunt; other implanted medical device (eg, insulin pump); metal fragments or foreign objects in the eyes, skin, or body; claustrophobia that would contraindicate a brain MRI scan
29. Brain MRI findings (or historical radiologic reports, if available) that show evidence of clinically significant structural brain disease which, in the opinion of the investigator, contraindicates performance of LP
30. Any spinal abnormality or other aspects (eg, tattoos) or other clinical findings (papilledema seen with ophthalmoscopy) that may complicate or contraindicate LP, as judged by the investigator
31. Ophthalmic abnormalities. The following are considered exclusionary:

    1. Congenital or acquired ophthalmic conditions (primary or secondary) that are considered poorly controlled within the last 12 months prior to screening, with or without treatment, or otherwise expected to lead to significant deterioration in visual acuity in the next 6 months after randomization
    2. Specific ophthalmic conditions:

    i. Current or past history of inflammation affecting the uveal tract or sclera ii. Diabetic retinopathy iii. Neovascular or exudative (wet) form of age-related macular degeneration iv. Active central serous retinopathy (central serous chorioretinopathy) v. Subjects with active autoimmune disease vi. Subjects taking immunosuppressive drugs (other than low doses of systemic steroids [< 10 mg per day of prednisone equivalent], for autoimmune disease that is considered to be inactive, in remission, or otherwise well-controlled). Other immunosuppressive drugs are contraindicated.

    vii. Mature cataracts (Grade ≥ 4 per the Lens Opacities Classification System III) or lower grade cataracts that are otherwise considered by the examining ophthalmologist to prevent adequate examination of the uveal tract or posterior ocular segment. (Note: Previous cataract surgery or an age-related cataract with age-appropriate lens opacification and no other important identified secondary causes [eg, diabetes, corticosteroids, vitamin deficiencies, trauma, radiation, or systemic fluid and electrolyte disturbances] is not necessarily exclusionary.)
32. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) concentrations >1.5 × the upper limit of normal (ULN) at screening, or between screening and baseline
33. Estimated creatinine clearance < 50 mL/min or creatinine > 1.5 × ULN at screening
34. Clinically significant vital sign abnormalities at screening or on Day 1, defined as (a) systolic blood pressure ≥ 160 mmHg, (b) diastolic blood pressure ≥ 90 mmHg (blood pressure assessed at rest; may be repeated up to 3 times), or (c) pulse rate < 45 or > 100 beats per minute (at rest)
35. Clinically significant abnormality in ECG rhythm, conduction or morphology at screening or between screening and randomization, including but not limited to:

    * Clinically significant PR (PQ) interval prolongation (PR > 220 msec)
    * Intermittent second or third degree atrioventricular (AV) block (AV block II Mobitz Type I, Wenckebach, while asleep or in deep rest is not exclusionary)
    * Bundle branch block or intraventricular conduction delay with QRS interval duration ≥ 120 msec
    * A Fridericia's corrected QT (QTcF) interval measurement > 470 msec, or a shortened QTcF < 340 msec, at screening or between screening and randomization; or a family history of long or short QT syndrome
36. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies, with relevant confirmatory testing conducted, where applicable, in accordance with Centers for Disease Control and Prevention guidance for HIV and viral hepatitis
37. Current blood clotting or bleeding disorder, including clinically significant abnormal findings in laboratory tests of coagulation
38. Poor venous access, such that IV drug delivery or PK/safety blood sampling would be difficult
39. Donation of blood or plasma within 2 months prior to screening and until 2 months after the final follow-up visit
40. A positive serum pregnancy test result at screening or prior to randomization
41. Urine drug screen positive for a drug of abuse (except for permitted, prescribed opiates and /or benzodiazepines). A urine drug screen positive for cannabinoids is exclusionary unless there is a documented legitimate medical reason for the subject's cannabinoid use (eg, chronic pain) or the investigator and medical monitor agree that the subject can abstain from use for the duration of the study.
42. Current employment by the sponsor (AstraZeneca) or by a contract research organization or clinical study site participating in this study, or a first-degree relative of an AstraZeneca employee or of an employee at a participating contract research organization or clinical study site

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 weeks
  Incidence, Nature, Severity and Seriousness of adverse events from screening
Vital Signs | 21 weeks
  Change from baseline in Blood Pressure measured in millimetres of Mercury
Oral Body Temperature | 21 weeks
  Change from baseline in body temperature measured in degrees Celcius
Body Weight | 21 weeks
  Change from baseline measured in Kilograms
Safety Laboratory Tests | 21 weeks
  Incidence from baseline in abnormal laboratory test results
Electrocardiograms | 21 weeks
  Change from baseline in ECG rythm
Ophthalmic assessments | 21 weeks
  Incidence from baseline in abnormal ocular findings
Suicidal Ideation | 21 weeks
  Evaluation of presence or absence of suicidal ideation as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
Cognitive impairment | 21 weeks
  Change from baseline in the total score of the Montreal Cognitive assessment; a 30-point test (the higher the score, the better the cognition)
Electrocardiograms | 21 weeks
  Change from baseline in ECG heart rate
Electrocardiograms | 21 weeks
  Change from baseline in ECG conduction
Electrocardiograms | 21 weeks
  Change from baseline in ECG PR interval
Electrocardiograms | 21 weeks
  Change from baseline in ECG QRS interval
Electrocardiograms | 21 weeks
  Change from baseline in ECG RR interval
Electrocardiograms | 21 weeks
  Change from baseline in ECG QT interval
Electrocardiograms | 21 weeks
  Change from baseline in ECG QTcF interval
Suicidal Behaviour | 21 weeks
  Evaluation of presence or absence of suicidal behaviour as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Beth E. Safirstein, MD, Principal Investigator — MD Clinical
Locations (5):
- United States (5):
  - Research Site, Long Beach, California
  - Research Site, Hallandale, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Farmington Hills, Michigan
  - Research Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymised individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de- identified individual patient-level data in an approved sponsor tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home